CLINICAL TRIAL: NCT01994629
Title: A Phase 2, Randomized, Controlled, Observer-Blind, Multi-Center Study Assessing the Safety and Immunogenicity of One Dose of Novartis' Meningococcal ACWY-CRM Vaccine and GlaxoSmithKline Biologicals' Meningococcal ACWY-TT Vaccine in Healthy Toddlers
Brief Title: Safety and Immunogenicity of One Dose of Novartis' Meningococcal ACWY-CRM Vaccine and GlaxoSmithKline Biologicals' Meningococcal ACWY-TT Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V59_67; 2013-000862-13 (EudraCT Number)
Record Dates: First submitted 2013-11-11; First posted 2013-11-26 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Meningococcal Disease
Keywords: meningococcal disease; children; vaccination
MeSH Terms: conditions — Meningococcal Infections | interventions — MenACWY-CRM vaccine; tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MenACWY-CRM (Experimental): MenACWY-CRM
  Interventions: Biological: MenACWY-CRM
- MenACWY-TT (Active Comparator): MenACWY-TT
  Interventions: Biological: MenACWY-TT

INTERVENTIONS:
Biological: MenACWY-CRM — MenACWY-CRM
  Arms: MenACWY-CRM
Biological: MenACWY-TT — MenACWY-TT
  Arms: MenACWY-TT

SUMMARY:
Evaluate the immune response and reactogenicity of one dose of Meningococcal ACWY-cross reactive material (CRM) and Meningococcal ACWY-tetanus toxoid (TT) in 12-15 months old healthy toddlers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children between 12 months and 15 months old inclusive who were born with an estimated gestational age ≥ 37 weeks.
2. Parent(s)/legal guardian(s) had given written informed consent after the nature of the study had been explained according to local regulatory requirements.
3. Parents/legal guardian available for all the visits and would comply with the requirements of the protocol (e.g., completion of the Diary Cards, availability for study visits / safety phone calls).
4. In good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. Previous confirmed or suspected disease caused by N. meningitidis.
2. Previously exposed to clinically proven meningococcal disease or clinical bacterial meningitis without further microbiologic characterization, i.e. possible meningococcal disease.
3. Previously immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s) (licensed or investigational).
4. Received within 90 days prior to enrollment or were expected to receive during the study period any investigational or non-registered product (drug or vaccine).
5. Received or planning to receive any vaccines within 14 days before and 30 days after administration of the study vaccine (Exceptions: Injectable influenza vaccine could be administered up to 14 days prior to study vaccination and at least 14 days after study vaccination).
6. Major congenital defect or a serious chronic disease.
7. History of any anaphylaxis, severe vaccine reactions, or allergy to any vaccine components including diphtheria toxoid (CRM197) or tetanus toxoid (TT) and latex.
8. Required chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the study vaccination. (For corticosteroids, this means prednisone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids were allowed).
9. Receipt of immunoglobulins and/or any blood products within six months prior to study vaccination or who had administration planned during the study period.
10. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
11. Any bleeding disorder which was considered as a contraindication to intramuscular injection.
12. Moderate or severe acute infection and/or fever (defined as temperature ≥ 38°C) within 3 days prior to enrollment.
13. Systemic antibiotic treatment within 7 days prior to enrollment.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (4):
- Italy (4):
  - Dipartimento di Prevenzione S C Igiene e Sanita Pubblica, Chiavari, ASL4 Chiavarese Regione Liguria Corso Dante 163
  - Ospedale Maggiore della Carita, Novara, Corso Mazzini 18
  - ASL Sassari 1 Servizio Igiene Pubblica, Sassari, Via Amendola 55
  - AOU Meyer Dip Scienze per la Salute della Donna e Bambino, Florence, Viale Pieraccini 24

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 4 centers in Italy.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- MenACWY-CRM (12 to 15 Months Old): Subjects received one dose of investigational MenACWY-cross reactive material (CRM) vaccine.
- MenACWY-TT (12 to 15 Months Old): Subjects received one dose of comparator MenACWY-tetanus toxoid (TT) vaccine.
Period: Overall Study
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Started | 100 | 102
Completed | 99 | 99
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- MenACWY-CRM (12 to 15 Months Old): Subjects received one dose of investigational MenACWY-CRM vaccine.
- MenACWY-TT (12 to 15 Months Old): Subjects received one dose of comparator MenACWY-TT vaccine.
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old) | Total
Number analyzed (Participants) | 100 | 102 | 202
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.8 (1) | 12.7 (0.9) | 12.7 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 94
  Male | 52 | 56 | 108
Region of Enrollment [Number; unit: Subjects]
  Italy | 100 | 102 | 202

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Severe Solicited Adverse Event (AE) After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT.
Description: Reactogenicity of MenACWY-CRM and comparator MenACWY-TT vaccine was assessed in subjects (12 to 15 months old) as measured by number of subjects with at least one severe solicited AE within 7 days after vaccination. Solicited AEs included tenderness, erythema, induration, irritability, sleepiness, change in eating habits, vomiting, diarrhea and fever.
Time Frame: Day 1 to Day 7 post-vaccination
Population: Analysis was done on the solicited safety data set (all subjects in the exposed set who provided post vaccination reactogenicity data: MenACWY-CRM 99; MenACWY-TT 101).
Measure: Number; unit: Number of Subjects
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 99 | 101
Number of Subjects | 4 | 2

2. Secondary Outcome: Percentages of Subjects With Human Serum Bactericidal Assay (hSBA) Titer ≥ 8 Against (N. Meningitidis) Serogroups A, C, W, and Y After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Immunogenicity of one dose of MenACWY-CRM and comparator MenACWY-TT vaccine was assessed in subjects (12 to 15 months old) as measured by the percentages of subjects with hSBA titer ≥ 8 directed against Neisseria meningitidis (N. meningitidis) serogroups A, C, W, and Y on Day 29 after vaccination. Persistence of immune responses was measured by the percentages of subjects with hSBA titer ≥ 8 on Day 180 post-vaccination.
Time Frame: Day 1, Day 29 and Day 180 post-vaccination
Population: Analysis was done on Full Analysis Set (FAS) Day 29 (subjects who received the vaccine and provided immunogenicity data at Day 29: MenACWY-CRM 95; MenACWT-TT 97). Persistence of immune responses at Day 180 was analysed on FAS Day 180 (subjects who received the vaccine and provided immunogenicity data at Day 180: MenACWY-CRM 98; MenACWT-TT 97).
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 98 | 97
percentage of Subjects
  A Day 1 (N=89,92) | 2 [0.27 to 7.9] | 0 [0 to 3.9]
  A Day 29 (N=91,97) | 90 [82.1 to 95.4] | 88 [79.4 to 93.4]
  A Day 180 (N=97,96) | 65 [54.6 to 74.4] | 30 [21.3 to 40.4]
  C Day 1 (N=92,93) | 3 [0.7 to 9.2] | 1 [0.03 to 5.8]
  C Day 29 (N=94,97) | 96 [89.5 to 98.8] | 86 [77 to 91.9]
  C Day 180 (N=96,95) | 88 [79.2 to 93.4] | 95 [88.1 to 98.3]
  W Day 1 (N=81,78) | 6 [2 to 13.8] | 4 [0.8 to 10.8]
  W Day 29 (N=84,87) | 62 [50.7 to 72.3] | 72 [61.8 to 81.5]
  W Day 180 (N=88,89) | 88 [78.7 to 93.6] | 100 [95.9 to 100]
  Y Day 1 (N=84,84) | 4 [0.7 to 10.1] | 2 [0.29 to 8.3]
  Y Day 29 (N=87,91) | 41 [30.9 to 52.4] | 56 [45.2 to 66.4]
  Y Day 180 (N=92,95) | 78 [68.4 to 86.2] | 98 [92.6 to 99.74]

3. Secondary Outcome: Percentages of Subjects With Seroresponse Against N. Meningitidis Serogroups A, C, W, and Y After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Immunogenicity of one dose of MenACWY-CRM and comparator MenACWY-TT vaccine was assessed in subjects (12 to 15 months old) as measured by the percentages of subjects with seroresponse defined as for subjects with pre-vaccination hSBA titer < 4, post-vaccination hSBA titer ≥ 8; for subjects with pre-vaccination hSBA titer ≥ 4, an increase of at least four times the pre-vaccination hSBA directed against N. meningitidis serogroups A, C, W, and Y on Day 29 after vaccination. Persistence immune response was measured by the percentage of subjects with seroresponse at Day 180 after vaccination.
Time Frame: Day 29 and Day 180 post-vaccination
Population: Analysis at Day 29 was done on FAS set at Visit Day 29. Persistence of immune responses at Day 180 was analysed on FAS at Visit Day 180.
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 98 | 97
percentage of Subjects
  A Day 29 (N=89,92) | 88 [79 to 93.7] | 87 [78.3 to 93.1]
  A Day 180 (N=95,92) | 62 [51.6 to 71.9] | 29 [20.3 to 39.8]
  C Day 29 (N=92,93) | 95 [87.8 to 98.2] | 84 [74.8 to 90.7]
  C Day 180 (N=94,92) | 85 [76.3 to 91.6] | 93 [86.3 to 97.6]
  W Day 29 (N=81,78) | 54 [42.9 to 65.4] | 73 [61.8 to 82.5]
  W Day 180 (N=83,81) | 83 [73.3 to 90.5] | 99 [93.3 to 99.97]
  Y Day 29 (N=84,84) | 39 [28.8 to 50.5] | 54 [42.4 to 64.5]
  Y Day 180 (N=88,87) | 74 [63.4 to 82.7] | 95 [88.6 to 98.7]

4. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against N. Meningitidis Serogroups A, C, W, and Y After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Immunogenicity of one dose of MenACWY-CRM and comparator MenACWY-TT vaccine was assessed in subjects (12 to 15 months old) as measured by hSBA GMTs directed against N. meningitidis serogroups A, C, W, and Y on Day 29 after vaccination. Persistence of immune response was measured by hSBA GMTs at Day 180 after vaccination.
Time Frame: Day 1, Day 29 and Day 180 post-vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 98 | 97
Titers
  A Day 1 (N=89,92) | 2.19 [2.02 to 2.38] | 2.04 [1.89 to 2.21]
  A Day 29 (N=91,97) | 41 [31 to 55] | 30 [23 to 40]
  A Day 180 (N=97,96) | 13 [9.5 to 18] | 4.67 [3.43 to 6.36]
  C Day 1 (N=92,93) | 2.44 [2.16 to 2.76] | 2.24 [1.99 to 2.52]
  C Day 29 (N=94,97) | 30 [23 to 39] | 20 [16 to 26]
  C Day 180 (N=96,95) | 24 [18 to 30] | 41 [32 to 53]
  W Day 1 (N=81,78) | 2.58 [2.12 to 3.15] | 2.4 [1.96 to 2.95]
  W Day 29 (N=84,87) | 9.34 [6.72 to 13] | 14 [9.91 to 19]
  W Day 180 (N=88,89) | 21 [17 to 27] | 56 [45 to 70]
  Y Day 1 (N=84,84) | 2.23 [2.02 to 2.48] | 2.16 [1.94 to 2.40]
  Y Day 29 (N=87,91) | 5.89 [4.27 to 8.13] | 8.20 [5.96 to 11]
  Y Day 180 (N=92,95) | 16 [12 to 21] | 26 [20 to 34]

5. Secondary Outcome: Percentages of Subjects With Rabbit Serum Bactericidal Assay (rSBA) Titer ≥ 8 Against Serogroups A, C, W, and Y After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Immunogenicity of one dose of MenACWY-CRM and comparator MenACWY-TT vaccine was assessed in subjects (12 to 15 months old) as measured by the percentages of subjects with rSBA titer ≥ 8 directed against N. meningitidis serogroups A, C, W, and Y on Day 29 after vaccination. Persistence of immune response was measured by percentages of subjects with rSBA titer ≥ 8 on Day 180 after vaccination.
Time Frame: Day 1, Day 29 and Day 180 post-vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 98 | 97
percentage of Subjects
  A Day 1 (rabbit; N=63,61) | 24 [14 to 36.2] | 31 [19.9 to 44.3]
  A Day 29 (rabbit; N=73,74) | 100 [95.1 to 100] | 100 [95.1 to 100]
  A Day 180 (rabbit; N=74,75) | 100 [95.1 to 100] | 93 [85.1 to 97.8]
  C Day 1 (rabbit; N=64,62) | 3 [0.38 to 10.8] | 0 [0 to 5.8]
  C Day 29 (rabbit; N=74,74) | 92 [83.2 to 97] | 97 [90.6 to 99.67]
  C Day 180 (rabbit; N=77,76) | 64 [51.9 to 74.3] | 71 [59.5 to 80.9]
  W Day 1 (rabbit; N=61,57) | 7 [1.8 to 15.9] | 5 [1.1 to 14.6]
  W Day 29 (rabbit; N=70,69) | 90 [80.5 to 95.9] | 91 [82 to 96.7]
  W Day 180 (rabbit; N=73,70) | 71 [59.4 to 81.2] | 87 [77 to 93.9]
  Y Day 1 (rabbit; N=61,59) | 10 [3.7 to 20.2] | 15 [7.2 to 27]
  Y Day 29 (rabbit; N=70,70) | 90 [80.5 to 95.9] | 89 [78.7 to 94.9]
  Y Day 180 (rabbit; N=74,71) | 80 [68.8 to 88.2] | 82 [70.7 to 89.9]

6. Secondary Outcome: Percentages of Subjects With rSBA Titer ≥ 128 Against Serogroups A, C, W, and Y After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Immunogenicity of one dose of MenACWY-CRM and comparator MenACWY-TT vaccine was assessed in subjects (12 to 15 months old) as measured by the percentages of subjects with rSBA titer ≥ 128 directed against N. meningitidis serogroups A, C, W, and Y on Day 29 after vaccination. Persistence of immune response was measured by percentages of subjects with rSBA titer ≥ 128 on Day 180 after vaccination.
Time Frame: Day 1, Day 29 and Day 180 post-vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 98 | 97
percentage of Subjects
  A Day 1 (rabbit; N=63,61) | 22 [12.7 to 34.5] | 31 [19.9 to 44.3]
  A Day 29 (rabbit; N=73,74) | 100 [95.1 to 100] | 100 [95.1 to 100]
  A Day 180 (rabbit; N=74,75) | 100 [95.1 to 100] | 91 [81.7 to 96.2]
  C Day 1 (rabbit; N=64,62) | 3 [0.38 to 10.8] | 0 [0 to 5.8]
  C Day 29 (rabbit; N=74,74) | 78 [67.3 to 87.1] | 65 [52.9 to 75.6]
  C Day 180 (rabbit; N=77,76) | 25 [15.6 to 35.8] | 33 [22.5 to 44.6]
  W Day 1 (rabbit; N=61,57) | 7 [1.8 to 15.9] | 5 [1.1 to 14.6]
  W Day 29 (rabbit; N=70,69) | 90 [80.5 to 95.9] | 90 [80.2 to 95.8]
  W Day 180 (rabbit; N=73,70) | 62 [49.5 to 72.8] | 66 [53.4 to 76.7]
  Y Day 1 (rabbit; N=61,59) | 10 [3.7 to 20.2] | 12 [4.9 to 22.9]
  Y Day 29 (rabbit; N=70,70) | 89 [78.7 to 94.9] | 86 [75.3 to 92.9]
  Y Day 180 (rabbit; N=74,71) | 73 [61.4 to 82.6] | 62 [49.7 to 73.2]

7. Secondary Outcome: Percentages of Subjects With Four-fold Increase in rSBA Titers Against Serogroups A, C, W, and Y After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Immunogenicity of one dose of MenACWY-CRM and comparator MenACWY-TT vaccine was assessed in subjects (12 to 15 months old) as measured by the percentages of subjects with four-fold increase in rSBA titer directed against N. meningitides serogroups A, C, W, and Y on Day 29 after vaccination. Persistence of immune response was measured by the percentages of subjects with four-fold increase in rSBA titer on Day 180 after vaccination.
Time Frame: Day 29 and Day 180 post-vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 98 | 97
percentage of Subjects
  A Day 29 (rabbit; N=63,61) | 100 [94.3 to 100] | 93 [84.1 to 98.2]
  A Day 180 (rabbit; N=60,61) | 97 [88.5 to 99.59] | 84 [71.9 to 91.8]
  C Day 29 (rabbit; N=64,62) | 75 [62.6 to 85] | 65 [51.3 to 76.3]
  C Day 180 (rabbit; N=64,63) | 20 [11.3 to 32.2] | 30 [19.2 to 43]
  W Day 29 (rabbit; N=61,57) | 87 [75.8 to 94.2] | 89 [78.5 to 96]
  W Day 180 (rabbit; N=58,58) | 55 [41.5 to 68.3] | 66 [51.9 to 77.5]
  Y Day 29 (rabbit; N=61,59) | 87 [75.8 to 94.2] | 88 [77.1 to 95.1]
  Y Day 180 (rabbit; N=61,59) | 72 [59.2 to 82.9] | 56 [42.4 to 68.8]

8. Secondary Outcome: rSBA GMT Against N. Meningitidis Against Serogroups A, C, W, and Y After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Immunogenicity of one dose of MenACWY-CRM and comparator MenACWY-TT vaccine was assessed in subjects (12 to 15 months old) as measured by rSBA GMTs directed against N. meningitidis serogroups A, C, W, and Y on Day 29 after vaccination. Persistence of immune responses was measured by rSBA GMTs on Day 180.
Time Frame: Day 1, Day 29 and Day 180 post-vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 98 | 97
Titers
  A Day 1 (rabbit; N=63,61) | 6.62 [3.12 to 14] | 12 [5.59 to 26]
  A Day 29 (rabbit; N=73,74) | 5698 [4226 to 7684] | 2827 [2116 to 3775]
  A Day 180 (rabbit; N=74,75) | 2815 [1741 to 4550] | 950 [592 to 1523]
  C Day 1 (rabbit; N=64,62) | 2.46 [1.98 to 3.05] | 2.07 [1.66 to 2.58]
  C Day 29 (rabbit; N=74,74) | 171 [113 to 259] | 142 [95 to 213]
  C Day 180 (rabbit; N=77,76) | 20 [12 to 33] | 22 [13 to 36]
  W Day 1 (rabbit; N=61,57) | 3.1 [2.09 to 4.59] | 3.17 [2.07 to 4.86]
  W Day 29 (rabbit; N=70,69) | 1092 [570 to 2089] | 1060 [553 to 2031]
  W Day 180 (rabbit; N=73,70) | 91 [46 to 182] | 142 [72 to 282]
  Y Day 1 (rabbit; N=61,59) | 3.46 [2.03 to 5.89] | 4.22 [2.42 to 7.38]
  Y Day 29 (rabbit; N=70,70) | 756 [400 to 1429] | 624 [333 to 1168]
  Y Day 180 (rabbit; N=74,71) | 248 [124 to 495] | 140 [70 to 278]

9. Secondary Outcome: Number of Subjects Reporting Solicited Adverse Events (AEs) After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Safety was assessed in terms of number of subjects (12 to 15 months old) reporting any and each of solicited local and systemic AEs reported from Day 1 to 7 after vaccination with one dose of either MenACWY-CRM or comparator MenACWY-TT vaccine.
Time Frame: Day 1 (6 hours) to Day 7 post-vaccination
Population: Analysis was done on solicited safety data set. MedDRA version v.3.0 was used for the analyses (in the AEs section, MedDRA version v.17.01 was used, leading to a different terminology to describe some of the events reported in this outcome).
Measure: Number; unit: Subjects
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 99 | 101
Subjects
  Any Local | 34 | 29
  Tenderness (N=97,100) | 29 | 26
  Erythema (N=97,100) | 4 | 2
  Induration (N=97,101) | 6 | 4
  Any Systemic | 56 | 57
  Irritability (N=96,99) | 30 | 39
  Sleepiness (N=96,98) | 23 | 26
  Change in eating habits (N=96,100) | 22 | 26
  Vomiting (N=96,99) | 6 | 9
  Diarrhea (N=96,99) | 17 | 18
  Fever (≥ 38.0°C; N=99,100)) | 14 | 13
  Prophylatic use of analg./antipyr. (N=97,100) | 1 | 4
  Therapeutic use of analg./antipyr. (N=98,100) | 13 | 13

10. Secondary Outcome: Number of Subjects Reporting Unsolicited (AEs) After Receiving One Dose of Either MenACWY-CRM Vaccine or MenACWY-TT Vaccine.
Description: Safety was assessed in terms of number of subjects (12 to 15 months old) reporting unsolicited AEs (day 1 to day 29), SAEs, medically attended AEs, AEs leading to premature study withdrawal (Day 1 to Day 180) after vaccination with one dose of either MenACWY-CRM or comparator MenACWY-TT vaccine.
Time Frame: Day 1 to Day 29 or Day 1 to Day 180 post-vaccination
Population: Analysis was done on unsolicited safety data set ie, all subjects in the exposed set who had post-vaccination unsolicited adverse event records.
Measure: Number; unit: Subjects
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Number analyzed (Participants) | 99 | 101
Subjects
  Any unsolicited AEs | 73 | 71
  AEs leading to premature withdrawal | 0 | 0
  SAEs | 8 | 3
  Medically attended AEs | 73 | 68
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 to Day 7 post vaccination, unsolicited AEs were collected from Day 1 to Day 29 post vaccination and SAEs, medically attended AEs and AEs leading to premature withdrawal were collected from Day 1 to Day 180.
Arm/Group | MenACWY-CRM (12 to 15 Months Old) | MenACWY-TT (12 to 15 Months Old)
Serious Adverse Events (participants affected / at risk) | 8/99 | 3/101
Other Adverse Events (participants affected / at risk) | 83/99 | 87/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM (12 to 15 Months Old) (N=99) | MenACWY-TT (12 to 15 Months Old) (N=101)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM (12 to 15 Months Old) (N=99) | MenACWY-TT (12 to 15 Months Old) (N=101)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (12)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 8 (8)
Somnolence (Nervous system disorders) | 23 (26) | 27 (30)
Injection site induration (General disorders) | 25 (26) | 26 (26)
Injection site pain (General disorders) | 29 (30) | 27 (27)
Pyrexia (General disorders) | 31 (44) | 34 (48)
Injection site erythema (General disorders) | 26 (26) | 27 (27)
Eating disorder (Psychiatric disorders) | 22 (27) | 26 (28)
Irritability (Psychiatric disorders) | 30 (37) | 40 (46)
Vomiting (Gastrointestinal disorders) | 8 (10) | 11 (13)
Diarrhea (Gastrointestinal disorders) | 21 (26) | 22 (29)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Conjunctivitis (Infections and infestations) | 6 (7) | 8 (9)
Ear infection (Infections and infestations) | 15 (20) | 4 (4)
Rhinitis (Infections and infestations) | 5 (5) | 2 (2)
Exhantema subitum (Infections and infestations) | 7 (7) | 5 (5)
Gastroenteritis (Infections and infestations) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other